CLINICAL TRIAL: NCT06248190
Title: Effectiveness of a Health Systems Strengthening Intervention to Improve Detection, Treatment, and Control of Multiple Long-Term Conditions in Primary Health Care Facilities in the Western Cape and KwaZulu Natal, South Africa
Brief Title: ENHANCE-EvideNce Led Co-created HeAlth Systems interventioNs for MLTCs CarE
Acronym: ENHANCE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of KwaZulu (Other)
Collaborators: University of Cape Town (Other); King's College London (Other); University of East Anglia (Other); University of Oxford (Other); Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Inge Petersen, Director, Centre for Rural Health, University of KwaZulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 686/2022; 201816 (Other Grant/Funding Number: NIHR); BREC/00005033/2022 (Other: UKZN BREC)
Record Dates: First submitted 2024-01-17; First posted 2024-02-08 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections; Hypertension; Diabetes Mellitus; Asthma; Depression; Myocardial Infarction; Stroke
Keywords: Multiple Chronic Conditions; Person Centered Care; Health Systems Intervention
MeSH Terms: conditions — HIV Infections; Hypertension; Diabetes Mellitus; Asthma; Depression; Myocardial Infarction; Stroke; Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: This study will be a type 2 hybrid trial, testing the effect of the intervention in improving clinical outcomes, and also testing and observing the effects of the intervention on implementation processes and outcomes using the RE-AIM (reach, effectiveness, adoption, implementation, maintenance) framework. The trial will be a cluster randomised parallel arm trial with embedded process evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): 1. Treatment literacy in chronic condition waiting rooms/pick-up points (posters, health promotion talks)
  2. 1-2 longer consultations with ENHANCE guide trained clinician
  3. Treatment literacy event - a contact between a CHW and a person with MLTC in their home (hopefully with carer), at 2 weeks and 4 weeks, using Health Diary
  4. Referrals to additional adherence counselling if necessary
  Interventions: Other: ENHANCE intervention (health systems)
- Control (No Intervention): Usual care at primary health care clinic, which includes consultation with a clinician using the PACK/APC guide. No additional support is usually provided for care of MLTCs.

INTERVENTIONS:
Other: ENHANCE intervention (health systems) — The intervention tools include a consolidated clinical decision support tool, health education posters, waiting room talks, medication list for treatment literacy and a patient health diary. Training session are delivered at all intervention sites and include 1 facility team session to introduce the ENHANCE study to the whole team; 3 clinical sessions for nurses and doctors; 2 sessions for community health workers and health promoters; Maintenance sessions to keep the ENHANCE intervention going for at least 12 months
  Arms: Intervention

SUMMARY:
The goal of this study is to determine the effect of the ENHANCE intervention in improving clinical outcomes and evaluating the effects of the intervention on implementation processes and outcomes. The specific questions it aims to answer are:

1. To test and estimate the effect of the intervention in people with MLTCs attending

   PHCs on:

   i. Detection of, and initiation of treatment for, additional chronic conditions ii. Treatment intensification and changes in medication iii. Control of chronic conditions iv. patient reported health-related quality of life and functioning v. health care utilisation and adherence vi. costs of health care
2. To use the RE-AIM framework to assess implementation processes and outcomes through measurements of reach, adoption, implementation, and maintenance.
3. To understand implementation processes and outcomes within the wider context of primary healthcare, provide explanations for the observed effects of the clinical findings and identify recommendations for wider implementation of the ENHANCE intervention.

The participants in the control group will receive usual care at their primary health care facility, which includes the use of the Practical Approach to Care Kit (PACK) or Adult Primary Care (APC) clinical decision support tool. Participants in the intervention group will receive care for their multiple chronic condition by a clinician trained to use the ENHANCE clinical decision support tool (intervention tool), and receive two CHW visits in their home to provide treatment literacy and adherence support.

DETAILED DESCRIPTION:
Control facilities Participants in control facilities will continue to receive usual care. Primary health care of long-term conditions is delivered free-at-point-of-care in public sector primary care facilities which includes the management of HIV, NCDs and mental health problems, according to South Africa's Ideal Clinic and Integrated Clinical Services Management model. This care model, which has combined the long-term care of HIV together with NCDs within each facility, has greatly enabled the feasibility of further interventions specifically addressing MLTCs and includes the Adult Primary Care (APC) or PACK clinical guidance. Patients attending these chronic services usually attend the same clinic regularly, 3 to 6-monthly for periodic monitoring of their chronic conditions. Chronic medication is collected monthly either at the facility (through fast-track queues), or through decentralised chronic medication dispensing systems which provide for collection from a range of sites including community venues (e.g. halls), wellness or adherence clubs, trailers, retail pharmacies (in KZN) or e-Lockers.

Intervention clinics

Participants in intervention clinics will continue with usual care as described for control clinics but in addition will receive the ENHANCE health systems intervention comprising tools and implementation strategies that have been co-developed with stakeholders through an iterative process, drawing on:

i. Evidence on the commonest MLTC combinations ii. Scoping reviews conducted on effectiveness of MLTCS interventions and systems barriers and enablers of person-centred care for MLTCs in LMICs iii. Provincial and district learning collaborative workshops with stakeholders from KZN and Western Cape.

iv. Clinical working groups with clinicians and health workers, a Guidance Oversight Board v. Input from our ENHANCE advocacy academy of 16 people living with MLTCs in the Western Cape and KZN

The intervention targets screening and early identification of other chronic conditions; improving follow-up and support for people with a new diagnosis, at risk of treatment failure (e.g. poorly controlled HIV or diabetes), and strengthen bi-directional referral pathways between the facility and community. Tools and implementation strategies will be layered into existing architecture of the chronic care system and support provision of more person-centred and empowering care across the treatment cascade.

Tools to support the implementation of the health systems intervention comprise:

* An integrated clinical decision support tool for care of MLTCs drawing on PACK/ APC.
* A range of patient-focussed materials to support condition, treatment, and systems (care-seeking) literacy (e.g., medication list, posters, scripts for health education talks)
* A personal health diary (paper-based)

Implementation strategies include:

* 1 facility team session to introduce the ENHANCE study to the whole team
* 3 clinical sessions for nurses and doctors
* 2 sessions for community health workers and health promoters
* Maintenance sessions to keep the ENHANCE intervention going for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 years and older
* At least two of the following conditions:

  i. HIV (Self-reported current treatment). ii. hypertension (Self-reported current treatment. iii. diabetes (Self-reported current treatment). iv. asthma, (Self-reported current treatment). vi. depression (Self-reported current treatment). vii. previous myocardial infarction (self-reported). viii. previous stroke (self-reported history).

Exclusion Criteria:

* Participants planning to relocate from either uMgungundlovu KwaZulu Natal and Cape Metro in Western Cape or changing their facilities during the period of the study.
* Participants who are unable to give informed consent due to loss of capacity.
* Participants self-reporting pregnancy
* Participants who cannot communicate in English, isiXhosa, isiZulu, or Afrikaans.
* Participants who are not willing to receive care for chronic conditions in their homes.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1837 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis and initiation of treatment during follow-up of one or more additional chronic condition | 12 months
  Number of participants with diagnosis of an additional chronic condition during follow-up (determined from medical records)
Intensification or change of treatment during follow-up for at least one of the chronic conditions present at enrolment. | 12 months
  Number of patients with increase in number of medication or doses or additional medications during the follow up period (determined by capturing of prescriptions at all visits)
Improved control of at least one condition that was not optimally controlled at baseline | 12 months
  This will include:HIV - viral suppression (viral load <50 copies/mL); hypertension - SBP/DBP<140 /90mmHg; diabetes - HbA1c <8%, Asthma Control Test score >16, Depression PHQ8 <10

SECONDARY OUTCOMES:
Functioning | 12 months
  A generic outcome of the primary outcome disaggregated by functioning (WHODAS-2.0)
Health-related quality of life | 12 months
  A generic outcome of the primary outcome disaggregated by health related quality of life (EQ-5D)
Adherence | 12 months
  A generic outcome of the primary outcome disaggregated by adherence (VAS)
Patient Experience of care | 12 months
  A generic outcome of the primary outcome disaggregated by patient experience of care (PACIC)
Depressive symptoms | 12 months
  A generic outcome of the primary outcome disaggregated by depressive symptoms (PHQ-8)
Patient experience with treatment and self-management | 12 months
  A generic outcome of the primary outcome disaggregated by patient experience with treatment and self-management (PETS)
Heathcare utilisation and cost | 12 months
  Health Utilisation and cost questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Helen Schneider, PhD, Study Chair — University of the Western Cape
Locations (32):
- South Africa (32):
  - Eastwood Clinic, Pietermaritzburg, KwaZulu-Natal
  - Esigodini Clinic, Pietermaritzburg, KwaZulu-Natal
  - Gcumisa Clinic, Pietermaritzburg, KwaZulu-Natal
  - Gomane Clinic, Pietermaritzburg, KwaZulu-Natal
  - Howick Clinic, Pietermaritzburg, KwaZulu-Natal
  - Impilwenhle Clinic, Pietermaritzburg, KwaZulu-Natal
  - Injabulo Clinic, Pietermaritzburg, KwaZulu-Natal
  - Mafatini Clinic, Pietermaritzburg, KwaZulu-Natal
  - Mphophomeni Clinic, Pietermaritzburg, KwaZulu-Natal
  - Ndaleni Clinic, Pietermaritzburg, KwaZulu-Natal
  - Northdale Clinic, Pietermaritzburg, KwaZulu-Natal
  - Pata Clinic, Pietermaritzburg, KwaZulu-Natal
  - Richmond Clinic, Pietermaritzburg, KwaZulu-Natal
  - Songonzima Clinic, Pietermaritzburg, KwaZulu-Natal
  - Willowfontein CHC, Pietermaritzburg, KwaZulu-Natal
  - Delft CHC, Cape Town, Western Cape
  - Dr Abdurahman CHC, Cape Town, Western Cape
  - DuNoon CHC, Cape Town, Western Cape
  - Durbanville CHC, Cape Town, Western Cape
  - Elsies CHC, Cape Town, Western Cape
  - Gugulethu CHC, Cape Town, Western Cape
  - Gustrouw CDC, Cape Town, Western Cape
  - Hanover Park CHC, Cape Town, Western Cape
  - Heideveld CHC, Cape Town, Western Cape
  - Kleinvlei CHC, Cape Town, Western Cape
  - Kraaifontein CHC, Cape Town, Western Cape
  - Macassar CDC, Cape Town, Western Cape
  - Michael M, Cape Town, Western Cape
  - Mitchells Plain CHC, Cape Town, Western Cape
  - Retreat CHC, Cape Town, Western Cape
  - Vanguard CHC, Cape Town, Western Cape
  - Caluza Clinic, Pietermaritzburg

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Background] Peer N, Uthman OA, Kengne AP. Rising prevalence, and improved but suboptimal management, of hypertension in South Africa: A comparison of two national surveys. Glob Epidemiol. 2021 Sep 10;3:100063. doi: 10.1016/j.gloepi.2021.100063. eCollection 2021 Nov. PMID 37635713
- [Background] Nguyen H, Manolova G, Daskalopoulou C, Vitoratou S, Prince M, Prina AM. Prevalence of multimorbidity in community settings: A systematic review and meta-analysis of observational studies. J Comorb. 2019 Aug 22;9:2235042X19870934. doi: 10.1177/2235042X19870934. eCollection 2019 Jan-Dec. PMID 31489279
- [Background] Hurst JR, Dickhaus J, Maulik PK, Miranda JJ, Pastakia SD, Soriano JB, Siddharthan T, Vedanthan R; GACD Multi-Morbidity Working Group. Global Alliance for Chronic Disease researchers' statement on multimorbidity. Lancet Glob Health. 2018 Dec;6(12):e1270-e1271. doi: 10.1016/S2214-109X(18)30391-7. No abstract available. PMID 30420026
- [Background] Mayosi BM, Flisher AJ, Lalloo UG, Sitas F, Tollman SM, Bradshaw D. The burden of non-communicable diseases in South Africa. Lancet. 2009 Sep 12;374(9693):934-47. doi: 10.1016/S0140-6736(09)61087-4. Epub 2009 Aug 24. PMID 19709736
- [Background] Oni T, Youngblood E, Boulle A, McGrath N, Wilkinson RJ, Levitt NS. Patterns of HIV, TB, and non-communicable disease multi-morbidity in peri-urban South Africa- a cross sectional study. BMC Infect Dis. 2015 Jan 17;15:20. doi: 10.1186/s12879-015-0750-1. PMID 25595711
- [Background] Gouda HN, Charlson F, Sorsdahl K, Ahmadzada S, Ferrari AJ, Erskine H, Leung J, Santamauro D, Lund C, Aminde LN, Mayosi BM, Kengne AP, Harris M, Achoki T, Wiysonge CS, Stein DJ, Whiteford H. Burden of non-communicable diseases in sub-Saharan Africa, 1990-2017: results from the Global Burden of Disease Study 2017. Lancet Glob Health. 2019 Oct;7(10):e1375-e1387. doi: 10.1016/S2214-109X(19)30374-2. PMID 31537368
- [Background] Kamkuemah M, Gausi B, Oni T. Missed opportunities for NCD multimorbidity prevention in adolescents and youth living with HIV in urban South Africa. BMC Public Health. 2020 Jun 1;20(1):821. doi: 10.1186/s12889-020-08921-0. PMID 32487118
- [Background] Herman AA, Stein DJ, Seedat S, Heeringa SG, Moomal H, Williams DR. The South African Stress and Health (SASH) study: 12-month and lifetime prevalence of common mental disorders. S Afr Med J. 2009 May;99(5 Pt 2):339-44. PMID 19588796
- [Background] COVID-19 Mental Disorders Collaborators. Global prevalence and burden of depressive and anxiety disorders in 204 countries and territories in 2020 due to the COVID-19 pandemic. Lancet. 2021 Nov 6;398(10312):1700-1712. doi: 10.1016/S0140-6736(21)02143-7. Epub 2021 Oct 8. PMID 34634250
- [Background] Roomaney RA, van Wyk B, Turawa EB, Pillay-van Wyk V. Multimorbidity in South Africa: a systematic review of prevalence studies. BMJ Open. 2021 Oct 6;11(10):e048676. doi: 10.1136/bmjopen-2021-048676. PMID 34615675